CLINICAL TRIAL: NCT04422639
Title: A Phase II Pilot Trial of Preoperative SRS/SRT Versus Postoperative SRS/SRT for Brain Metastases
Brief Title: Preoperative SRS/SRT vs Postoperative SRS/SRT for Brain Metastases
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Following the EAB for NCI Designation this study was identified as having no funding and not meeting enrollment goals. It was requested by the EAB that this study be closed due to inactivity.
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 260505
Record Dates: First submitted 2020-05-29; First posted 2020-06-09 (Actual); Results first posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm I (pre-operative SRS/SRT) (Experimental): Patients undergo SRS or SRT within 15 days of randomization followed by surgery within 15 days of radiation completion. Patients may undergo additional SRS or SRT if disease returns after treatment.
  Interventions: Radiation: SRS/SRT
- Arm II (post-operative SRS/SRT) (Active Comparator): Patients undergo surgery within 15 days of randomization followed by standard-of-care SRS or SRT within 30 days of surgery. Patients may undergo additional SRS or SRT if disease returns after treatment.
  Interventions: Radiation: SRS/SRT

INTERVENTIONS:
Radiation: SRS/SRT — Comparing pre-operative SRS/SRT to post-operative SRS/SRT

SUMMARY:
This pilot study is a randomized, open-label, 2-arm active-controlled phase II clinical trial conducted at a single study site (UAMS). Subjects will be randomized to one of the 2 treatment arms and stratified by size of index lesion and number of brain metastases.

The investigators will prospectively compare preoperative (neoadjuvant) SRS/SRT to postoperative (adjuvant) SRS/SRT in patients undergoing surgical resection for brain metastases.

The investigators hypothesize that neoadjuvant SRS/SRT prior to surgical resection of brain metastases will result in improved freedom from Central Nervous System (CNS) events when compared to adjuvant SRS/SRT after surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prior histopathological diagnosis of cancer other than small cell lung cancer, lymphoma, and germ cell histologies.
* MR imaging of the brain with findings strongly suggestive of metastatic tumor(s) as assessed by the radiologist.
* Seen by a neurosurgeon or radiation oncologist and judged to be appropriate for participation in this study, including the ability to tolerate both surgery and SRS/SRT, e.g., the ability to lie flat in a stereotactic soft head frame.
* ECOG ≤ 2
* 1-2 index lesion(s) appropriate for resection, not previously treated with SRS/SRT.

Index lesion(s) should be > 2 cm and < 5 cm in largest dimension, and require resection. Alternatively, patients with a diagnosis of melanoma and a lesion < 1.5cm in largest dimension may also be included. o All other brain lesions must be appropriate for SRS/SRT alone and treated according to physician preference. Prior neurosurgery and/or prior SRS/SRT at a non-overlapping location are permitted at the discretion of the treating physician.

- MRI confirmed 1-10 lesions, 1-2 of which are the index lesions undergoing surgery.

Each non-index lesion (up to 10) must measure ≤ 3.0 cm in maximal extent on contrasted MRI scan, and not otherwise require resection.

* Clinical indication and plan for stereotactic radiosurgery to all known brain lesions requiring treatment (≤ 10 metastases).
* Surgical resection able to be performed within 15 days of radiotherapy completion.
* Written informed consent obtained from subject, or a legally designated power of attorney and ability for subject to comply with the requirements of the study.
* Negative pregnancy test in women of childbearing potential (WOCBP) within 30 days of radiation. WOCBP is a female patient less than 50 years of age or who has menstruated within the last 12 months.
* Platelet count > 80 k/cumm, Hgb > 7.5 gm/dL, INR < 1.3, ANC > 1.5 k/cumm

Exclusion Criteria:

* Not a surgical candidate per neurosurgeon's discretion.
* Contraindication to general anesthesia.
* Not a radiosurgical candidate per radiation oncologist's discretion.
* Metastatic germ cell tumor, small cell carcinoma, leukemia, multiple myeloma or lymphoma or any primary brain tumor
* ECOG > 2
* < 3 months expected survival
* Radiologic documentation of hydrocephalus in addition to symptoms of hydrocephalus
* Radiographic or cytologic evidence of leptomeningeal disease.
* Imaging Findings:

  * Midline shift > 6mm
  * >10 lesions, one of which is the index lesion
  * Largest lesion > 5cm
* Pregnancy
* Known allergy to gadolinium, pacemaker, or other contraindication such as metal implant that is not safe for MRI. Patients with MRI-compatible implants are eligible.
* Patients who have local recurrence of previously treated brain metastasis.
* Patients who have received prior WBRT.
* Inherited radiation hypersensitivity syndromes

  o Ataxia Telangiectasia, Nijmegen Breakage Syndrome, Fanconi Anemia, DNA Ligase IV, Mre 11 deficiency, SCID, Bloom's syndrome
* Collagen vascular diseases

  o Active systemic lupus erythematous (SLE), scleroderma, mixed connective tissue disorder, polymyositis or dermatomyositis, CREST Syndrome
* Cytotoxic Chemotherapy within 7 days prior to SRS/SRT.

  o Molecularly targeted therapies, including immune-modulatory drugs, can be given within 7 days of SRS/SRT at the discretion of the treating physician.
* Patients who received anti-VEGF therapy within 6 weeks prior to enrollment, as there is increased risk of fatal brain hemorrhage with surgical resection.
* Treatment plan respecting normal tissue tolerances using dose fractionation specified within the protocol cannot be achieved.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Analiz Rodriguez, MD, PhD, Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Pre-operative SRS/SRT) | Arm II (Post-operative SRS/SRT)
Started | 1 | 2
Completed | 0 | 0
Not Completed | 1 | 2
Not completed — Death | 1 | 0
Not completed — study closed prior to completion of FU visits | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Pre-operative SRS/SRT) | Arm II (Post-operative SRS/SRT) | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Central Nervous System (CNS) Composite Event (CE)
Description: A CNS CE will consist of one of the following three events: Local Recurrence (LR) of the treated lesions, symptomatic radiation necrosis (SRN) to the treated lesions, or development of leptomeningeal disease (LMD).
Time Frame: From date of randomization to the date of a documented LR, SRN, or LMD, whichever comes first, assessed up to 18 months.
Population: No data displayed because Outcome Measure has zero total participants analyzed due to low enrollment and early study termination. Study closed prior to completion of follow-up visits so there is nothing to analyze.
Arm/Group | Arm I (Pre-operative SRS/SRT) | Arm II (Post-operative SRS/SRT)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Arm I (Pre-operative SRS/SRT) | Arm II (Post-operative SRS/SRT)
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/2
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Pre-operative SRS/SRT) (N=1) | Arm II (Post-operative SRS/SRT) (N=2)
Left hemiplegia (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Pre-operative SRS/SRT) (N=1) | Arm II (Post-operative SRS/SRT) (N=2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Vision decrease (Eye disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Edema cerebral (Nervous system disorders) | 0 (0) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Outcome measures not computed because study closed prior to completion of follow-up visits so there is nothing to analyze.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/39/NCT04422639/Prot_SAP_000.pdf